CLINICAL TRIAL: NCT04390529
Title: A Multicenter, Observational Cohort Study of Women Undergoing Immediate Breast Reconstruction Following MAstectomy (IRMA)
Brief Title: Immediate Breast Reconstruction Following Mastectomy (IRMA)
Acronym: IRMA
Status: Active, not recruiting | Type: Observational
Sponsor: Thurgau Breast Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRMA
Record Dates: First submitted 2020-04-27; First posted 2020-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quality-of-life questionnaire: BREAST-Q — quality-of-life questionnaire: BREAST-Q

SUMMARY:
Based on data from the US Surveillance, Epidemiology and End Result Program (SEER), the rates of nipple-sparing mastectomy (NSM) have risen 202% since 2009. In spite of the increasing popularity of IRMA, limited research has been done to identify complications in patients undergoing these procedures. Of particular importance is to assess the effects of combining the procedure with radiotherapy, and undergoing a one- versus two-step surgical procedure.

Active monitoring and periodic assessment of IRMA patients are needed to establish the safety of these different techniques in terms of complications and recurrence rates. Identifying an optimal strategy for IRMA may lead to the development of clinical guidelines, which are currently lacking.

DETAILED DESCRIPTION:
This is a multicenter observational, cohort study. The study is designed to serve a similar purpose as a disease registry. The only study-specific intervention will be the completion of the BREAST-Q quality-of-life (QoL) form. Only quantitative data will be collected. The rationale for this study design is to identify and describe the type and frequency of complications related to IRMA. No hypothesis is being tested. Although group comparisons based on surgical techniques will be made, conclusions based on these findings will be limited by the observational nature of the design.

Data from patients will be collected using a series of pseudonymized case report forms, including the validated quality-of-life questionnaire: BREAST-Q. These data will be entered into the web-based data collection system, SecuTrial. A precise description of the surgical procedure will be required, as specified on the case report forms (e.g., implantation of a mesh, resection margins), to allow for subsequent multivariate analyses.

During the first year of follow-up, data from routine clinical assessments and the QoL forms will be gathered at baseline (within 90 days after mastectomy), 6 and 12 months. Thereafter, data will be collected from annual clinical assessments and completion of the QoL form will be done for an additional four years (24, 36, 48 and 60 months postoperatively). Consequently, a total of five years of postoperative follow-up data will be collected to allow sufficient time for the development of the majority of foreseeable complications.

ELIGIBILITY:
Inclusion Criteria:

* Any women ≥ 18 years of age undergoing IRMA (NSM or SSM) at any participating breast center may be included in the study.
* Women undergoing IRMA for either prophylactic or oncologic purposes
* Enrolment is possible up to 90 days after mastectomy
* A patient who has had the mastectomy at a non-participating institution, but has subsequently sought treatment at one of the study centers, may be eligible for enrolment up to 90 days following mastectomy

Exclusion Criteria:

* Unwillingness to have follow-up assessments at the participating breast centers
* Limited ability to understand study-specific procedures, which includes language difficulties.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Study Population: Women undergoing IRMA (NSM: nipple-areola sparing mastectomy or SSM: skin-sparing mastectomy) at any participating breast center may be included in the study. Patients undergoing IRMA for either prophylactic or oncologic purposes are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of nipple-areola complex (NAC) or skin flap necrosis requiring specific treatment/surgery | Three years after surgery
  Postoperative follow-up assessments include the documentation of nipple-areola complex (NAC) or skin flap necrosis
Rate of infection requiring surgery | Three years after surgery
  Postoperative follow-up assessments include the documentation of infections requiring surgery
Grade of surgical complications | Three years after surgery
  Postoperative follow-up assessments include the documentation of surgical complications (grading according to Clavien-Dindo Classification of Surgical Complications)

SECONDARY OUTCOMES:
Rate of minor complications not requiring surgery | Three years after surgery
  Postoperative follow-up assessments include the documentation of skin necrosis outside NAC, wound dehiscence, and seroma requiring drainage
Level of patient satisfaction with cosmesis | Five years after surgery
  Postoperative follow-up assessment using BREAST-Q quality-of-life questionnaire that measures patient satisfaction with cosmetic outcome
Level of sensitivity of the operated breast (NAC) compared to the non-operated breast | Five years after surgery
  Postoperative follow-up assessments of breast functional outcomes
Rate of breast cancer recurrence | Five years after surgery
  Postoperative follow-up assessments include the documentation of recurrence in the NAC, skin flap outside the NAC, chest wall, locoregional lymph node (axillary, supraclavicular), distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Fehr, Prof. Dr., Principal Investigator — Brustzentrum Thurgau, Spital Thurgau AG
Locations (15):
- Switzerland (15):
  - Kantonsspital Aarau AG, Aarau, Canton of Aargau
  - Kantonsspital Baden, Prof. Dr. med. Cornelia Leo, Baden, Canton of Aargau
  - Brustzentrum Bern Biel, Hirslanden, Bern, Canton of Bern
  - Centre du Sein de Genève - Hirslanden Clinique des Grangettes, Chêne-Bougeries, Canton of Geneva
  - Tumor- und Brustzentrum ZeTuP, Sankt Gallen, Canton of St. Gallen
  - Brustzentrum Ostschweiz, Sankt Gallen, Canton of St. Gallen
  - Tumor- und BrustZentrum Ostschweiz, Sankt Gallen, Canton of St. Gallen
  - Spital Wetzikon, Wetzikon, Canton of Zurich
  - Brust Centrum Zürich, Bethanien & Zollikerberg, Zollikerberg, Canton of Zurich
  - Stadtspital Triemli, Zurich, Canton of Zurich
  - Ente Ospedaliero Cantonale (Ospedale Regionale di Bellinzona e Valli and Ospedale Regionale di Lugano), Lugano, Canton Ticino
  - Brustzentrum Thurgau, Spital Thurgau AG, Prof. Dr. med. Mathias K. Fehr, Frauenfeld, Thurgau
  - Campus SLB Sonnenhof AG, Bern
  - HUG - Hôpitaux universitaires de Genève, Geneva
  - Universitätsspital Zürich, Klinik für Gynäkologie, Zurich

IPD SHARING:
Plan to Share IPD: No